CLINICAL TRIAL: NCT00966238
Title: A Phase II, Open-label, Escalating Dose-ranging Study to Evaluate the Safety and Immunogenicity of VAX125 Influenza Vaccine in Community-living Adults ≥65 Years of Age
Brief Title: Safety and Immunogenicity of VAX125 Influenza Vaccine in Community-living Adults >= 65 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VaxInnate Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VAX125-02
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Results first posted 2011-07-14 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Influenza
Keywords: influenza; vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VAX125 (Experimental): HA1 influenza vaccine
  Interventions: Biological: VAX125

INTERVENTIONS:
Biological: VAX125 — STF2.HA1(SI) (VAX125), which is a recombinant fusion protein that consists of Salmonella typhimurium flagellin type 2 (STF2), a Toll-like receptor 5 (TLR5) ligand, fused at its C-terminus to the globular head domain of the hemagglutinin (HA) antigen of influenza A HA1 Solomon Islands (SI).

SUMMARY:
A multi-center, open-label, escalating dose-ranging study to assess the safety, reactogenicity, and immunogenicity of four different VAX125 vaccine doses; 0.5 µg, 1.0 µg, 2.0 µg, or 3.0 µg, delivered i.m. as a single dose vaccination on Day 0. Hypothesis: VAX125 is safe and immunogenic at one or more of the doses tested.

DETAILED DESCRIPTION:
A total of 80 community-living adults who are ≥65 years of age will be enrolled across the four dose groups. Following vaccination, each subject will remain at the study site for at least 30 minutes to be observed for any immediate reactogenicity complaints associated with the Day 0 vaccination. Subjects will also be evaluated during clinic visits on Study Days 1, 7, 14, and 28 following vaccination. In addition, a safety follow-up telephone contact will occur on post vaccination Day 3.

There will be 20 subjects per dose group. Up to 3 study sites will enroll 6-10 subjects per dose group over a two-day enrollment period. Progression to the next higher dose group will take place only if the Safety Monitoring Committee (SMC) assessment of the 30 (+15) minutes, Day 0, and Day 1 post vaccination safety data; Day 3 telephone report: and the Day 0 and Day 1 serum C-reactive protein (CRP) results concludes that the lower dose was well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women aged 65 or older; female subjects must be post menopausal.
* Live in the community, independently or in an assisted living environment
* Based on the results of the Short Portable Mental Status Questionnaire (SPMSQ), be rated as normal or have no greater than mild severity dementia.
* As defined by the Canadian Study of Health and Aging Clinical Frailty Scale (CSHA-CFS), fitness ranging from very fit to mildly frail; Classes 1 to 5 of 7.
* Healthy volunteers, as determined by medical history, physical examination (PE), vital signs, and clinical safety laboratory examinations.
* Able to comprehend the study requirements, agree to its provisions, have the ability to adhere to the provisions of the study, and give written informed consent prior to study entry.
* Willing to receive the unlicensed (VAX125) vaccine given as an i.m. injection.
* Willing to provide multiple blood specimens collected by venipuncture.

Exclusion Criteria:

* Persons who in the opinion of the Investigator, have a psychiatric illness, a chronic illness (e.g., diabetes or liver or kidney disease), or who are taking a concomitant therapy or have any other condition that would interfere with the subject's participation in the study or interpretation of the study results.
* Persons having cancer or have received treatment for cancer within three years (persons with a history of cancer who are disease-free without treatment for three years or more are eligible.
* Persons with impaired immune responsiveness (of any cause), including diabetes mellitus.
* Persons presently receiving or having a recent history of receiving (within the past six months) any medication or therapeutic modality that affects the immune system such as allergy shots, immune globulin, interferon, immunomodulators, radiation therapy, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable). Inhaled and topical corticosteroids are allowed.
* Persons who have had a prior serious reaction to influenza vaccine.
* Persons with a history of anaphylactic-type reaction to injected vaccines.
* Persons with a history of drug or chemical abuse in the year prior to screening.
* Persons currently participating in another research study involving study medications (drugs or vaccines) or who have participated within 30 days of vaccination.
* Persons who have received blood or blood products within eight weeks prior to vaccination or are planning to receive blood or blood products during the study period.
* Persons who have donated blood or blood products within eight weeks prior to vaccination or plan to donate at any time during the study.
* Persons with acute disease within 72 hours prior to vaccination defined as the presence of a moderate or severe illness as determined by the Investigator through medical history and physical examination. Vaccination can be delayed until the subject has recovered.
* Persons with significant cardiovascular disease e.g., New York Heart Associate (NYHA) Class 3 or 4 congestive heart failure; myocardial infarction within the past six months; unstable angina, coronary angioplasty within the past six months; uncontrolled ventricular cardiac arrhythmias; resting heart rate (HR) >100 beats per minute (bpm)
* Persons with a history of chronic obstructive pulmonary disease or history of other lung disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Taylor, MD, Study Director — VaxInnate Corporation
Locations (3):
- United States (3):
  - JCCT, Lanexa, Kansas
  - Univ of Rochester, Rochester, New York
  - Coastal Carolina Research Center, Charleston, South Carolina

REFERENCES:
- [Derived] Taylor DN, Treanor JJ, Strout C, Johnson C, Fitzgerald T, Kavita U, Ozer K, Tussey L, Shaw A. Induction of a potent immune response in the elderly using the TLR-5 agonist, flagellin, with a recombinant hemagglutinin influenza-flagellin fusion vaccine (VAX125, STF2.HA1 SI). Vaccine. 2011 Jul 12;29(31):4897-902. doi: 10.1016/j.vaccine.2011.05.001. Epub 2011 May 17. PMID 21596084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 3 clinical sites.
Period: Overall Study
Arm/Group | 0.5 µg i.m. | 1.0 µg i.m. | 2.0 µg i.m. | 3.0 µg i.m. | 5.0 µg i.m. | 8.0 µg i.m.
Started | 20 | 20 | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 µg i.m. | 1.0 µg i.m. | 2.0 µg i.m. | 3.0 µg i.m. | 5.0 µg i.m. | 8.0 µg i.m. | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 20 | 20 | 20 | 20 | 20 | 20 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (6.12) | 71.2 (4.65) | 71.7 (4.16) | 71.9 (4.28) | 70.7 (4.07) | 70.6 (4.91) | 71.5 (4.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 10 | 5 | 12 | 9 | 53
  Male | 10 | 13 | 10 | 15 | 8 | 11 | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local and Systemic Immediate Reactogenicity Complaints
Time Frame: within 4 hours following vaccination
Population: Immediate complaints were vaccination symptoms that were solicited and observed at 30 minutes (+15 minutes) and (±30 minutes) after the vaccination on Day 0.
Measure: Number; unit: Participants
Arm/Group | 0.5 µg i.m. | 1.0 µg i.m. | 2.0 µg i.m. | 3.0 µg i.m. | 5.0 µg i.m. | 8.0 µg i.m.
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Participants
  Redness | 0 | 0 | 0 | 0 | 0 | 0
  Swelling | 0 | 0 | 0 | 0 | 0 | 0
  Bruising | 0 | 0 | 0 | 0 | 0 | 0
  Arm Pain | 8 | 8 | 6 | 7 | 9 | 11
  Headache | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue | 0 | 0 | 1 | 0 | 0 | 0
  Joint Pain | 0 | 0 | 0 | 0 | 1 | 1
  Muscle Aches | 0 | 0 | 1 | 0 | 2 | 1
  Chills | 0 | 0 | 0 | 0 | 0 | 0
  Sweating | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Geometric Mean Hemagglutinin Inhibition (HAI) Antibody Titers
Time Frame: 28 days after vaccination
Population: The immunogenicity of the vaccine was evaluated by measuring the number of subjects who demonstrate seroconversion either by developing a measurable titer following vaccination or by showing a significant increase in HAI serum antibody titers post-vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 0.5 µg i.m. | 1.0 µg i.m. | 2.0 µg i.m. | 3.0 µg i.m. | 5.0 µg i.m. | 8.0 µg i.m.
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Titers
  Baseline | 27.32 [14.34 to 52.04] | 27.32 [15.00 to 49.77] | 24.62 [11.87 to 51.09] | 50.98 [29.13 to 89.22] | 18.59 [10.01 to 34.53] | 30.31 [15.93 to 57.70]
  Day 7 | 30.31 [15.79 to 58.20] | 38.64 [21.21 to 70.39] | 50.98 [24.72 to 105.12] | 105.56 [49.64 to 224.50] | 66.66 [37.85 to 117.42] | 154.55 [85.63 to 278.94]
  Day 14 | 42.87 [22.05 to 83.35] | 77.27 [43.22 to 138.16] | 69.64 [33.95 to 142.86] | 160.00 [82.23 to 311.32] | 230.44 [119.96 to 442.68] | 234.25 [127.42 to 430.68]
  Day 28 | 47.57 [23.88 to 94.76] | 74.64 [44.15 to 126.21] | 69.64 [33.95 to 142.86] | 149.29 [78.77 to 282.93] | 222.18 [113.51 to 434.89] | 211.12 [120.49 to 369.94]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected for 1 year following vaccination. All adverse events were collected for 28 days following vaccination.
Arm/Group | 0.5 µg i.m. | 1.0 µg i.m. | 2.0 µg i.m. | 3.0 µg i.m. | 5.0 µg i.m. | 8.0 µg i.m.
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20 | 0/20 | 1/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 2/20 | 0/20 | 0/20 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 µg i.m. (N=20) | 1.0 µg i.m. (N=20) | 2.0 µg i.m. (N=20) | 3.0 µg i.m. (N=20) | 5.0 µg i.m. (N=20) | 8.0 µg i.m. (N=20)
Breast Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 µg i.m. (N=20) | 1.0 µg i.m. (N=20) | 2.0 µg i.m. (N=20) | 3.0 µg i.m. (N=20) | 5.0 µg i.m. (N=20) | 8.0 µg i.m. (N=20)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less